CLINICAL TRIAL: NCT05792579
Title: Early Versus Late Stoma Closure After Traumatic Colorectal Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahgoub Abd Elmonem Mahgoub, assiut, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Early and late stoma closure
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Stoma Colostomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early closure of stoma (Active Comparator): Detection complications of early closure of stoma in pateints with colorectal injures
  Interventions: Procedure: stoma closure
- late closure of stoma (Active Comparator): Detection complications of late closure of stoma.
  Interventions: Procedure: stoma closure

INTERVENTIONS:
Procedure: stoma closure — early closure of stoma in trauma patients

SUMMARY:
The aim is to study feasibility,advantages and disadvantages of early closure of stoma versus late closure of stoma

DETAILED DESCRIPTION:
Most traumatic colon injuries can be repaired primarily, but a stoma may still be required for severe colonic or rectal injury. The current trend is to reverse the stoma early, rather than to wait the traditional 3 months before closure)1-3) Trauma patients, however, are usually young and otherwise healthy individuals, with an excellent potential for optimal healing once they have overcome the initial insult. It is these patients who could benefit from early closure of the stoma(4-6). Once the temporary stoma has been constructed, various reasons have been cited for the development of colon-related complications after closure. The timing of the operation, the age of the patient, the type of colostomy, and the use of primary or delayed skin closure have all been implicated(7-8). Of all these, the timing of the operation is the most controversial. The early closure of a temporary stoma has many attractions. It can reduce hospitalization time and cost, eliminates the need for stoma care by the patient, and abolishes the psychologic, social, and financial burdens of a stoma in an otherwise healthy person(9-11)

ELIGIBILITY:
Inclusion Criteria:

* age between (10-50)

Exclusion Criteria:

* pathological causes
* deep, open perineal tear
* Severe co-morbid conditions (uncontrolled diabetes, Hypertension)

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Early versus late stoma closure after traumatic colorectal injuries | Baseline
  Detection complications of early closuare of stoma

REFERENCES:
- [Background] Taheri PA, Ferrara JJ, Johnson CE, Lamberson KA, Flint LM. A convincing case for primary repair of penetrating colon injuries. Am J Surg. 1993 Jul;166(1):39-44. doi: 10.1016/s0002-9610(05)80579-3. PMID 8328627
- [Background] Todd GJ, Kutcher LM, Markowitz AM. Factors influencing the complications of colostomy closure. Am J Surg. 1979 Jun;137(6):749-51. doi: 10.1016/0002-9610(79)90086-2. PMID 453467